CLINICAL TRIAL: NCT03011333
Title: A Phase 2B, Randomized, Controlled Study of HTX-011 Administered Via Pectoral Nerve Block in Subjects Undergoing Upper Extremity Surgery for Augmentation Mammoplasty
Brief Title: Phase 2B Upper Extremity Nerve Block Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTX-011-211
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group 1: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam), 60 mg/1.8 mg via nerve block.
  Interventions: Drug: HTX-011
- Group 2: HTX-011 (Experimental): HTX-011(bupivacaine/meloxicam), 120 mg/3.6 mg via nerve block.
  Interventions: Drug: HTX-011
- Group 3: HTX-011 (Experimental): HTX-011(bupivacaine/meloxicam), 240 mg/7.2 mg via nerve block.
  Interventions: Drug: HTX-011
- Group 4: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg via nerve block.
  Interventions: Drug: HTX-011
- Group 5: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam), 400 mg/ 12 mg via instillation.
  Interventions: Drug: HTX-011
- Group 6: Bupivacaine HCl (Active Comparator): Bupivacaine HCl without epinephrine, 50 mg via nerve block.
  Interventions: Drug: Bupivacaine HCl without epinephrine
- Group 7: Saline Placebo (Placebo Comparator): Saline placebo via nerve block.
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: HTX-011 — HTX-011 (bupivacaine/meloxicam) via nerve block or instillation.
  Arms: Group 1: HTX-011; Group 2: HTX-011; Group 3: HTX-011; Group 4: HTX-011; Group 5: HTX-011
Drug: Bupivacaine HCl without epinephrine — Bupivacaine HCl without epinephrine, 50 mg via nerve block.
  Arms: Group 6: Bupivacaine HCl
Drug: Saline Placebo — Saline placebo via nerve block.
  Arms: Group 7: Saline Placebo

SUMMARY:
This is a Phase 2B, randomized, assessor-blind, active- and saline placebo-controlled, multicenter study in subjects undergoing augmentation mammoplasty to evaluate the analgesic efficacy, safety, and pharmacokinetics (PK) of HTX-011 when administered via ultrasound-guided lateral and medial pectoral nerve block before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo primary bilateral submuscular augmentation mammoplasty with saline or silicone smooth implants with a volume of 300 to 500 cc, inclusive. Note: textured implants are not allowed.
* Has an American Society of Anesthesiologists Physical Status of I, II, or III.
* Subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Has a planned concurrent surgical procedure.
* Has a planned reconstructive procedure status post breast cancer therapy.
* Has a pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medication.
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken NSAIDs within 10 days prior to scheduled surgery.
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has been administered any local anesthetic within 72 hours prior to the scheduled surgery other than to treat an AE that occurs after signing the ICF or for pretreatment prior to a needle placement.
* Has initiated treatment with any of the following medications within 1 month prior to study drug administration or is taking any of these medications to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin, duloxetine, or cyclooxygenase-2 (COX-2) inhibitors. (Note: If a subject is taking one of these medications for a reason other than pain control, she must be on a stable scheduled dose [ie, not "as needed"] for at least 1 month prior to study drug administration.) Anxiolytics prior to surgery are permitted, if necessary.
* Has a medical condition that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* Has a known history of Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV).
* Has uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments
* Has any chronic neuromuscular deficit of either pectoral nerve function or arm/shoulder/truncal musculature.
* Has any chronic condition or disease that would compromise neurological or vascular assessments.
* Had a malignancy in the last year, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention-deficit/hyperactivity disorder, benzodiazepine for anxiety disorder) may be eligible for participation in the study. Subjects taking medical marijuana are not allowed to participate in the study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half lives.
* Has undergone 3 or more surgeries in 12 months.
* Has a body mass index (BMI) >35 kg/m2.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2017-01-14 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pasadena, California
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 243 subjects received study drug.
Period: Overall Study
Arm/Group | Group 1: HTX-011 | Group 2: HTX-011 | Group 3: HTX-011 | Group 4: HTX-011 | Group 5: HTX-011 | Group 6: Bupivacaine HCl | Group 7: Saline Placebo
Started | 12 | 27 | 25 | 47 | 50 | 41 | 41
Completed | 12 | 26 | 25 | 46 | 46 | 37 | 36
Not Completed | 0 | 1 | 0 | 1 | 4 | 4 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 4 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: HTX-011 | Group 2: HTX-011 | Group 3: HTX-011 | Group 4: HTX-011 | Group 5: HTX-011 | Group 6: Bupivacaine HCl | Group 7: Saline Placebo | Total
Number analyzed (Participants) | 12 | 27 | 25 | 47 | 50 | 41 | 41 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 27 | 25 | 47 | 50 | 41 | 41 | 243
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.4 (6.56) | 32.1 (8.51) | 30.5 (5.64) | 30.9 (8.08) | 32.0 (8.64) | 30.4 (7.75) | 31.3 (9.03) | 31.2 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 27 | 25 | 47 | 50 | 41 | 41 | 243
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 10 | 18 | 17 | 17 | 16 | 94
  Not Hispanic or Latino | 6 | 17 | 15 | 29 | 33 | 24 | 25 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 3 | 2 | 2 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 3 | 6 | 11 | 3 | 7 | 36
  White | 10 | 22 | 20 | 38 | 37 | 35 | 32 | 194
  More than one race | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 27 | 25 | 47 | 50 | 41 | 41 | 243

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores With Activity (NRS-A) Through 24 Hours Postsurgery (AUC0-24).
Description: Pain intensity is assessed using an 11-point NRS (0-10) where 0 represents "no pain" and 10 represents "worst pain imaginable" (using windowed worst observation carried forward to adjust for opioid rescue medication use). The theoretical range of AUC0-24 is 0-240. The prescribed activity for NRS-A is keeping the elbows at the side and against the body and then raising both hands in front of the abdomen with hands clasped and holding that position for at least 5 seconds.
Time Frame: 24 hours
Population: mITT Population
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Group 1: HTX-011 | Group 2: HTX-011 | Group 3: HTX-011 | Group 4: HTX-011 | Group 5: HTX-011 | Group 6: Bupivacaine HCl | Group 7: Saline Placebo
Number analyzed (Participants) | 12 | 27 | 25 | 12 | 50 | 41 | 41
pain intensity score*hr | 124.51 (59.462) | 136.17 (58.598) | 136.76 (56.034) | 116.71 (52.622) | 114.87 (48.214) | 133.83 (49.493) | 151.52 (46.213)

2. Secondary Outcome: Mean Total Postoperative Opioid Consumption (in Morphine Equivalents)
Time Frame: 72 Hours
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents (MME)
Arm/Group | Group 1: HTX-011 | Group 2: HTX-011 | Group 3: HTX-011 | Group 4: HTX-011 | Group 5: HTX-011 | Group 6: Bupivacaine HCl | Group 7: Saline Placebo
Number analyzed (Participants) | 12 | 27 | 25 | 47 | 50 | 41 | 41
Morphine milligram equivalents (MME) | 38.71 (28.650) | 24.39 (19.878) | 38.00 (19.452) | 28.84 (22.603) | 37.46 (21.452) | 33.57 (23.088) | 36.38 (23.275)

ADVERSE EVENTS:
Time Frame: 28 Days.
Description: Subjects reporting more than one Treatment Emergent Adverse Event (TEAE) are counted only once.
Arm/Group | Group 1: HTX-011 | Group 2: HTX-011 | Group 3: HTX-011 | Group 4: HTX-011 | Group 5: HTX-011 | Group 6: Bupivacaine HCl | Group 7: Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/27 | 0/25 | 0/47 | 0/50 | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/27 | 1/25 | 0/47 | 1/50 | 2/41 | 0/41
Other Adverse Events (participants affected / at risk) | 11/12 | 21/27 | 23/25 | 43/47 | 47/50 | 33/41 | 35/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: HTX-011 (N=12) | Group 2: HTX-011 (N=27) | Group 3: HTX-011 (N=25) | Group 4: HTX-011 (N=47) | Group 5: HTX-011 (N=50) | Group 6: Bupivacaine HCl (N=41) | Group 7: Saline Placebo (N=41)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: HTX-011 (N=12) | Group 2: HTX-011 (N=27) | Group 3: HTX-011 (N=25) | Group 4: HTX-011 (N=47) | Group 5: HTX-011 (N=50) | Group 6: Bupivacaine HCl (N=41) | Group 7: Saline Placebo (N=41)
Dizziness (Nervous system disorders) | 1 | 6 | 10 | 4 | 6 | 8 | 4
Headache (Nervous system disorders) | 0 | 4 | 4 | 3 | 7 | 4 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 5 | 5 | 2 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 5 | 6 | 2 | 2
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 2 | 2 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 6 | 6 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 15 | 14 | 37 | 37 | 25 | 26
Vomiting (Gastrointestinal disorders) | 4 | 6 | 7 | 17 | 19 | 14 | 16
Constipation (Gastrointestinal disorders) | 2 | 4 | 2 | 7 | 7 | 6 | 8
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 4 | 2 | 4 | 7 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 6 | 1 | 3 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 2 | 4 | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0 | 4 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 5 | 3 | 2 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 1 | 3 | 4 | 5 | 2 | 4
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 6 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT03011333/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03011333/SAP_001.pdf